CLINICAL TRIAL: NCT04113057
Title: Role of Provider Feedback in Home-based Walking Programs Utilizing Smart Devices
Brief Title: Home-based Walking Program With Smart Devices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In-person supervised exercise therapy (SET) at this institution, a required component of this study, was halted during Covid19 and was not re-instated after clinical activities resumed.
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shirling Tsai, Physician, Dallas VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-022
Record Dates: First submitted 2019-09-26; First posted 2019-10-02 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: PAD - Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: prospective randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Coaching (Experimental): All subjects enrolled in the study will be enrolled in supervised exercise therapy. They will also receive directions for supplemental home-based exercise and a LIVMOR remote health monitoring system. The remote coaching arm will receive regular provider feedback based on LIVMOR data.
  Interventions: Other: Remote Coaching
- Remote health monitoring without provider feedback (No Intervention): All subjects enrolled in the study will be enrolled in supervised exercise therapy. They will also receive directions for supplemental home-based exercise and a LIVMOR remote health monitoring system. The "no intervention" arm will have access to LIVMOR data, but without provider feedback on the LIVMOR data.

INTERVENTIONS:
Other: Remote Coaching — In patients randomized to the remote coaching arm, study staff will provide feedback on home-based supplemental exercise based on heart rate and walking distance measurements from the LIVMOR health monitoring system.
  Arms: Remote Coaching

SUMMARY:
Intermittent claudication (IC), the most common manifestation of peripheral artery disease (PAD), represents not only a significant detriment in quality of life, but also an increased risk for atherosclerotic cardiovascular disease (ASCVD), including progression of PAD, coronary artery disease (CAD) and cerebrovascular disease. Guideline directed therapy for IC includes supervised exercise, smoking cessation and optimal medical management to decrease overall risk of ASCVD. In the VA Health Care System, implementation of supervised exercise therapy through cardiac rehabilitation or physical therapy programs is limited by distances that patients must travel to VA facilities that provide these services. Furthermore, one of the most common failure points in exercise therapy programs is poor patient compliance. Improved patient participation and compliance in exercise programs for IC represents an unmet need, without which the majority of patients with life-style limiting PAD may not be receiving optimal medical management.

Small studies have demonstrated the effectiveness of home-based exercise programs as an alternative to supervised exercise therapy; however, the success of the home-based exercise programs require remote coaching and/or regular provider feedback. The wide-spread availability of smart phones and smart devices has accelerated the implementation of telehealth programs that may supplement or may eventually replace in-person encounters for health care delivery. The role of provider feedback in addition to real-time feedback from smart devices remains completely unexplored. Our central hypothesis is that in individuals with IC, regular provider feedback on smart-device-based remote health monitoring data, which is available to the patient in real time, will augment the benefits of home-based exercise programs. We propose a randomized trial in patients with IC to test the central hypothesis through two Specific Aims:

1. To determine the effect of provider feedback on smart-device-based remote health monitoring data during home-based exercise programs on walking distance in patients with IC.
2. To determine the effect of provider feedback on smart-device-based remote health monitoring data during home-based exercise programs on quality of life (QOL) in patients with IC.

Based on a sample size calculation to detect a 50% increase in walking distance between the 2 groups, we expect to enroll 30 patients (15 in each group). Patient participation in the study will be concluded after 12 weeks.

As an exploratory aim in the study, we will also (as an optional part of the study) collect plasma before and after the 12-weeks of exercise to investigate changes in lipid levels and plasma biomarkers associated with exercise therapy. This exploratory aim will generate preliminary data for future studies.

DETAILED DESCRIPTION:
The study design is that of a prospective randomized study of patients presenting to the vascular surgery and cardiology clinics with symptoms of IC and enrolled in 12-week supervised exercise program. Upon enrollment, each patient will undergo a medical and surgical history, ascertainment of smoking status, review of medications, and 6-minute walk test (walking on a flat, pre-defined course(i.e. hallway) for 6 minutes and recording time and distance to claudication onset as well as total distance walked, and total number of steps taken). We will also collect data from the patient's CPRS notes through our institutional cardiac rehab/PAD rehab program, with a dedicated cardiac rehab nurse. Patients with IC who are enrolled in the study will also be asked to complete 2 QOL questionnaires: the VASCUQoL6 and the Walking Impairment Questionnaire (WIQ). Patients will undergo supervised exercise therapy (per cardiac rehab protocol) and will receive the LIVMOR health monitoring system with instructions on how to use it. Randomization and details of exercise therapy are described in the next section. Patients will be followed for up to 12 weeks to collect data regarding change in distance and time of claudication onset.

In the optional exploratory aim, we will analyze plasma from one blood draw at the beginning and at the end of exercise therapy for lipid levels, distribution of LDL particle size, and other biomarkers. We will perform metabolomics, proteomics, and lipidomics assays to examine small circulating molecules that are involved in the development of atherosclerotic plaque in peripheral arterial disease. All blood and plasma analysis performed outside of Pathology and the Clinical Core Lab will be performed in the PI's research laboratory at the Dallas VA Medical Center by members of the research staff, or by members of the PI's collaborating lab at UT Southwestern or in the UT Southwestern research Core Laboratories. Any plasma sent to UT Southwestern will be de-identified.

Data (including name, birth date, social security number, dates of procedures and studies) will be stored in an Excel spreadsheet. Each patient's data will be associated with a study ID and stripped of the 18 identifiers need to de-identify the data. Only study staff will have access to PHI. No PHI will be released outside the North Texas VA Health Care Systems.

For the LIVMOR system, only the patient's study ID will be entered into the system. De-identified health monitoring data (heart rate, steps taken, distance walked) will be transmitted and stored in the LIVMOR cloud server, as was done in the LIVMOR Data Collection Study (IRB# 17-106).

After enrollment, baseline data, including questionnaires, will be collected. Patients who have agreed to optional blood draw will have a fasting blood draw (up to 10 cc) at the next available time within 1 week of study enrollment. At the next supervised exercise therapy visit (occurs 3 times a week according to the cardiac rehab protocol), the patient will have baseline resting heart rate and blood pressure measurements, and will undergo a 6-minute walk test. The patient will be randomized to remote coaching (regular provider feedback based on LIVMOR data) vs. remote health monitoring without provider feedback. Each patient will be sent home with instructions for home-based supplemental exercise and a LIVMOR remote health monitoring system, which includes a wristwatch that records heart rate, steps taken, and distance traveled (pedometer function) and a tablet. Patients will be instructed to check a resting heart rate with the LIVMOR watch for 10 minutes before starting exercise. They will exercise while wearing the watch (heart rate monitor and pedometer), then check heart rate for 10 minutes after completion of the exercise session. Patients will not receive real time feedback from the smart-watch heart rate monitor, however they have the option to review their heart rate and pedometer data by logging into the tablet provided with the watch, after the exercise session. In patients randomized to the remote coaching arm, study staff will provide feedback on home-based supplemental exercise based on heart rate measurements and pedometer measurements from the LIVMOR health monitoring system, as well as heart rate and walking data collected from supervised exercise therapy sessions. Remote coaching will occur by telephone call, but the conversation will mirror conversations that occur during supervised exercise therapy, and will not be based solely on the surrogate measure of heart rate for walking effort. A member of the study team will call the patient 1-3 times a week, depending on the patient's preference, which may change over the course of the study. Therefore the remote coaching is adaptive to patient's needs. In patients randomized to no remote coaching, health monitoring data will be reviewed by study staff, but will not be used to adjust home-based supplemental exercise. Any abnormalities in health monitoring data will be alerted to appropriate clinical staff. All patients will keep a journal of their home-based supplemental exercise, including time of exercise, in order to correlate heart rate readings from the smart-watch.

For patients agreeing to the optional blood draw: Blood will be sent to the Dallas VA Medical Center clinical lab for a lipid panel. The remaining blood will be refrigerated, then transported to the PI's research lab at the Dallas VA Medical Center, where the research staff will centrifuge the blood to isolate plasma.

Plasma will be tested for the following:

* Metabolomics, proteomics, and lipidomics assays to study small circulating molecules that may be involved in the development of atherosclerosis in peripheral arterial disease, and may change with exercise therapy.
* Lipoprotein subfractions.
* Small molecules that can be assayed using ELISA. At the end of the 12-week program, an end-of-study 6 minute walk test will be performed as well as the questionnaires will be completed. All the LIVMOR devices will be returned to the investigators. If the patient is unable to complete the end-of study 6-min walk test or does not complete the 12-week exercise program, a phone follow- up will be done to complete the questionnaires. A final blood draw will be completed (within 1 week of completing the 12-week exercise program) for patients who have opted for the blood draw.

The LIVMOR system transmits data through wireless technology up to a cloud server. The data transmission is encrypted and FIPS-140-2 compliant.

ELIGIBILITY:
Inclusion Criteria:

* Presence of documented PAD by ABI <0.90 at rest or ≥20% drop in claudication limited exercise ABI in either limb and one of the following criteria in the corresponding limb:

  i. Prior lower extremity revascularization ii. Known presence of flow-limiting stenosis (≥70%) by clinically indicated angiography, computed tomographic (CT) or magnetic resonance imaging (MRI), or Duplex ultrasonography (DUS)
* Documented diagnosis of intermittent claudication
* Enrollment in supervised exercise therapy through the institutional cardiac rehab program

Exclusion Criteria:

* Severe cardiac or pulmonary disease that precludes participation in an exercise-based study.
* Severe psychiatric or behavioral illness that precludes study participation
* Inability to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Maximal walking distance | Baseline to 12 weeks
  Change in distance to claudication onset (e.g. pain in the legs that limits walking)

SECONDARY OUTCOMES:
Change in Quality of life measured by the VASCUQoL6 | Baseline to 12 weeks.
  Change in quality of life as measured by the VASCUQoL6 Questionnaire
Change in Quality of life measured by the WIQ Questionnaire | Baseline to 12 weeks.
  Change in quality of life as measured by the WIQ Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas VAMC, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Background] Banerjee S, Sarode K, Vinas A, Banerjee A, Mohammad A, Brilakis ES. The role of antiplatelet therapy in patients with peripheral artery disease and lower extremity peripheral artery revascularization. Curr Opin Cardiol. 2015 Sep;30(5):525-35. doi: 10.1097/HCO.0000000000000208. PMID 26241710
- [Background] Bonaca MP, Scirica BM, Creager MA, Olin J, Bounameaux H, Dellborg M, Lamp JM, Murphy SA, Braunwald E, Morrow DA. Vorapaxar in patients with peripheral artery disease: results from TRA2degreesP-TIMI 50. Circulation. 2013 Apr 9;127(14):1522-9, 1529e1-6. doi: 10.1161/CIRCULATIONAHA.112.000679. Epub 2013 Mar 15. PMID 23501976
- [Background] Conn NJ, Schwarz KQ, Borkholder DA. In-Home Cardiovascular Monitoring System for Heart Failure: Comparative Study. JMIR Mhealth Uhealth. 2019 Jan 18;7(1):e12419. doi: 10.2196/12419. PMID 30664492
- [Background] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Background] Fakhry F, van de Luijtgaarden KM, Bax L, den Hoed PT, Hunink MG, Rouwet EV, Spronk S. Supervised walking therapy in patients with intermittent claudication. J Vasc Surg. 2012 Oct;56(4):1132-42. doi: 10.1016/j.jvs.2012.04.046. PMID 23026425
- [Background] Gardner AW, Parker DE, Montgomery PS, Blevins SM. Step-monitored home exercise improves ambulation, vascular function, and inflammation in symptomatic patients with peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2014 Sep 18;3(5):e001107. doi: 10.1161/JAHA.114.001107. PMID 25237048
- [Background] Gardner AW, Parker DE, Montgomery PS, Scott KJ, Blevins SM. Efficacy of quantified home-based exercise and supervised exercise in patients with intermittent claudication: a randomized controlled trial. Circulation. 2011 Feb 8;123(5):491-8. doi: 10.1161/CIRCULATIONAHA.110.963066. Epub 2011 Jan 24. PMID 21262997
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FGR, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RAG, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Mar 21;69(11):e71-e126. doi: 10.1016/j.jacc.2016.11.007. No abstract available. PMID 27851992
- [Background] Hageman D, Fokkenrood HJ, Gommans LN, van den Houten MM, Teijink JA. Supervised exercise therapy versus home-based exercise therapy versus walking advice for intermittent claudication. Cochrane Database Syst Rev. 2018 Apr 6;4(4):CD005263. doi: 10.1002/14651858.CD005263.pub4. PMID 29627967
- [Background] Harwood AE, Cayton T, Sarvanandan R, Lane R, Chetter I. A Review of the Potential Local Mechanisms by Which Exercise Improves Functional Outcomes in Intermittent Claudication. Ann Vasc Surg. 2016 Jan;30:312-20. doi: 10.1016/j.avsg.2015.05.043. Epub 2015 Sep 9. PMID 26362620
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] McDermott MM. Exercise training for intermittent claudication. J Vasc Surg. 2017 Nov;66(5):1612-1620. doi: 10.1016/j.jvs.2017.05.111. Epub 2017 Sep 2. PMID 28874320
- [Background] McDermott MM. Medical Management of Functional Impairment in Peripheral Artery Disease: A Review. Prog Cardiovasc Dis. 2018 Mar-Apr;60(6):586-592. doi: 10.1016/j.pcad.2018.03.007. Epub 2018 May 1. PMID 29727608
- [Background] McDermott MM, Guralnik JM, Criqui MH, Ferrucci L, Zhao L, Liu K, Domanchuk K, Spring B, Tian L, Kibbe M, Liao Y, Lloyd Jones D, Rejeski WJ. Home-based walking exercise in peripheral artery disease: 12-month follow-up of the GOALS randomized trial. J Am Heart Assoc. 2014 May 21;3(3):e000711. doi: 10.1161/JAHA.113.000711. PMID 24850615
- [Background] Montgomery PS, Gardner AW. The clinical utility of a six-minute walk test in peripheral arterial occlusive disease patients. J Am Geriatr Soc. 1998 Jun;46(6):706-11. doi: 10.1111/j.1532-5415.1998.tb03804.x. PMID 9625185
- [Background] Sood A, Watts SA, Johnson JK, Hirth S, Aron DC. Telemedicine consultation for patients with diabetes mellitus: a cluster randomised controlled trial. J Telemed Telecare. 2018 Jul;24(6):385-391. doi: 10.1177/1357633X17704346. Epub 2017 Apr 13. PMID 28406066
- [Background] Wang A. Review of vorapaxar for the prevention of atherothrombotic events. Expert Opin Pharmacother. 2015;16(16):2509-22. doi: 10.1517/14656566.2015.1099629. Epub 2015 Oct 19. PMID 26480240